CLINICAL TRIAL: NCT06306781
Title: Clinical Trial Evaluating the Efficacy of Homologous Allogeneic Hepatocytes in Patients With Decompensated Cirrhosis
Brief Title: A Clinical Trial Evaluating the Safety, Tolerability, and Preliminary Efficacy of HCL001 Cell Injection (Homologous Allogeneic Hepatocytes) in Patients With Decompensated Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HI-IM-002
Record Dates: First submitted 2024-01-31; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCL001 cell injection (homologous allogeneic hepatocytes) (Experimental): low/middle/high dose group
  Interventions: Drug: HCL001 cell (homologous allogeneic hepatocytes) injection

INTERVENTIONS:
Drug: HCL001 cell (homologous allogeneic hepatocytes) injection — The patient will undergo a DSA procedure in the hospital's operating room before infusion. A catheter will be inserted into the femoral artery and guided to the hepatic artery. Upon confirmation through imaging, HCL001 cell injection will be slowly infused through the catheter. During the infusion, the cells should be continuously agitated to prevent clumping. The infusion can be administered as a single dose or multiple doses, and after infusion, the patient will be closely monitored for at least one week.

SUMMARY:
This study protocol is designed to evaluate the clinical efficacy, safety, and tolerability of HCL001 cell injection in the treatment of decompensated cirrhosis. The aim is to provide stronger evidence for the clinical application of HCL001 cell injection in the treatment of decompensated cirrhosis, thereby attempting to improve patients' survival and quality of life to meet the clinical needs for treating decompensated liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* When signing the informed consent form, individuals between the ages of 18 to 75 years (inclusive, including the boundary values) are eligible, and there are no restrictions based on gender.
* According to the "Guidelines for the Diagnosis and Treatment of Cirrhosis (2019 Edition)", a diagnosis of decompensated cirrhosis is made.
* A Child-Pugh score of 7-12 points (including the threshold) is classified as [insert the corresponding classification as per the provided appendix].
* An ECOG performance status score of 0-2 or a Karnofsky Performance Status (KPS) score greater than 60 is considered [insert the corresponding classification or interpretation].
* A safe vascular access that allows for hepatic intra-arterial catheterization and angiography
* If screening for patients with hepatitis B or C-related cirrhosis, the viral load should be ≤1000 IU/mL for HBV-DNA and ≤15 IU/mL for HCV-RNA. For patients with alcoholic cirrhosis, the abstinence period should be ≥6 months.
* During screening, the serum ALT level should be ≤3 times the upper limit of normal (ULN).
* Understand and adhere to the research process, voluntarily participate, and sign the informed consent form (the informed consent form is to be voluntarily signed by myself or a legally authorized representative).

Exclusion Criteria:

* Allergic individuals, especially those allergic to any component of HCL001 cell injection or its excipients.
* Individuals with concurrent liver cancer or other malignant tumors.
* Patients who are unable or unwilling to cooperate or comply with the requirements of the research protocol.
* International Normalized Ratio (INR) >2.5 and platelet count (PLT) less than 30 x 10^9/L.
* Patients who have used anticoagulant or antiplatelet medications within the past week prior to screening.
* Patients with a history of upper gastrointestinal bleeding or spontaneous peritonitis within the past four weeks prior to screening.
* Patients who have experienced grade 3 or higher hepatic encephalopathy within the past three months prior to administering the medication.
* Patients with severe dysfunction in vital organs such as the heart, lungs, brain, or kidneys, including: History of severe lung diseases such as severe emphysema, pulmonary embolism, or other lung conditions that significantly impact lung function. Significant history of heart disease that meets either of the following conditions: a. Decompensated heart failure (New York Heart Association [NYHA] class III-IV). b. Unstable angina. Chronic kidney disease, such as chronic nephritis, renal insufficiency, or uremia.
* For patients with diabetes mellitus that is being treated but not effectively controlled, it typically refers to those with a glycated hemoglobin (HbA1c) level of ≥8%.
* Patients with severe coagulation dysfunction or bleeding disorders, such as hemophilia, as well as those with severe jaundice indicated by a serum total bilirubin level of ≥171 μmol/L.
* This includes pregnant or lactating women, as well as individuals who are unable or unwilling to follow the researcher's guidance in using the approved contraceptive measures during the study period and for 6 months after the study ends.
* Those who have received stem cell therapy in the past, or who are currently participating in another interventional clinical trial or have been enrolled in one within the past 3 months, are excluded from screening.
* HIV positive
* Presence of active infection during screening
* The researchers consider any other factors that are not suitable for trial inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Types and incidence of treatment-related adverse events. | The entire process of treatment (up to 48 weeks).
  Recording the types and incidence of treatment-related adverse events.
Dose-Limiting Toxicity (DLT) | 28 days after the completion of treatment.
  Recording the Dose-Limiting Toxicity (DLT) . If one or more instances of Dose-Limiting Toxicity (DLT) occur, the dose escalation according to the original plan will be stopped, and the previous dose level will be determined as the Maximum Tolerated Dose (MTD).
Maximum Tolerated Dose (MTD) | 28 days after the completion of treatment.
  Recording Maximum Tolerated Dose (MTD).If one or more instances of Dose-Limiting Toxicity (DLT) occur, the dose escalation according to the original plan will be stopped, and the previous dose level will be determined as the Maximum Tolerated Dose (MTD).

SECONDARY OUTCOMES:
Child-Pugh grading. | On the 7th day, 28th day, 42nd day (only for multiple-dose group), 56th day (only for multiple-dose
  Child-Pugh scoring is a scoring system used to assess the liver function and prognosis of patients with cirrhosis, typically used to evaluate the severity of liver disease in patients. Child-Pugh scoring is based on several indicators of the patient, including the following five indicators:
  Total bilirubin levels Albumin levels Coagulation function (prothrombin time or PT) Degree of Ascites Presence of hepatic encephalopathy Child-Pugh scoring assesses the above five indicators and classifies patients into three grades A, B, or C, representing mild, moderate, and severe conditions respectively. A higher score indicates more severe liver dysfunction.
  Child-Pugh scoring is primarily used to evaluate the liver function and prognosis of patients with liver disease, assisting physicians in developing treatment plans and assessing the severity of the patients' conditions.
Number of participants with abnormal laboratory tests results | On the 7th day, 28th day, 42nd day (only for multiple-dose group), 56th day (only for multiple-dose
  Objective laboratory tests/examinations (ALT, AST, TBIL, DBIL, TP, ALB, GLB, Hb, white blood cell count, and platelet count.)
The percentage of participants with improved liver conditions (including changes in portal vein diam | At week 12, 24, and 48 after the initial administration of medication.
  Ultrasound examination

IPD SHARING:
Plan to Share IPD: No